CLINICAL TRIAL: NCT02177045
Title: Breast Lesions Characterization on Contrast Enhanced Ultrasound With Histopathological Correlation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 0164-14-RMB CTIL
Record Dates: First submitted 2014-06-26; First posted 2014-06-27 (Estimated); Last update posted 2014-10-01 (Estimated); Status verified 2014-09

CONDITIONS: Malignant Neoplasm, Overlapping Lesion of Breast
MeSH Terms: conditions — Neoplasms | interventions — contrast agent BR1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Microbubbles contrast media for US (Experimental): Sonovue, Bracco, microbubbles contrast media
  Interventions: Drug: Sonovue, Bracco

INTERVENTIONS:
Drug: Sonovue, Bracco — Intravenous injection

SUMMARY:
Breast lesions are a common condition, diagnosed by imaging and palpation. In order to reduce the number of biopsies performed to the definitive diagnosis of a breast lesion, an imaging method with a high degree of accuracy is needed. Ultrasound imaging with microbubbles contrast media allows the diagnosis of vascularization of the lesion, according to timing. Our hypothesis is that a highly vascularized lesion that enhances in an early timing is most likely to represent a malignant lesion and thus, deserves biopsy for a definitive diagnosis. Females over 18 years age, with a focal lesion in breast will be suitable to perform this examination.

ELIGIBILITY:
Inclusion Criteria:

* Female with a diagnosed breast focal lesion

Exclusion Criteria:

* Allergic conditions to contrast media,
* asthma,
* R-L shunt

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2014-10; Primary Completion 2015-10 (Estimated); Study Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
Tumor vascularization | one year

CONTACTS AND LOCATIONS:
Overall Officials: Diana Gaitini, Prof, Principal Investigator — Rambam Health Care Center
Locations (1):
- Ultrasound Unit Imaging Dept Rambam Health Care Campus, Haifa, Israel